CLINICAL TRIAL: NCT01234584
Title: Soft and Hard Tissue Changes Around the New Lance® Implants Using Traditional and Switch Platform Abutments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr. zvi Gutmacher, Department of Maxillofacial Rehabilitation School of Gradute Dentistry Rambam Health care campus Haifa, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CTIL0227-10-RMB
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-09

CONDITIONS: Group A- 23 Implant Using Switch Platform -SPK Abutment.; Group B- 22 Implant Using the Traditional -CPK Abutment.
MeSH Terms: interventions — MAP Kinase Kinase 1

ARMS (2):
- Group A (Experimental): 23 implants using SPK Abutments
  Interventions: Procedure: spk
- Group B (Active Comparator): implants using CPK Abutments
  Interventions: Procedure: CPK Abutments

INTERVENTIONS:
Procedure: spk — implants using SPK Abutments
  Arms: Group A
Procedure: CPK Abutments — implants using CPK Abutments
  Arms: Group B

SUMMARY:
The purpose of this present study is to compare alveolar bone changes and markers of gingival health around the new Lanes® dental implant which were rehabilitate using the new switch platform abutment ( SPR ) and the traditional ( CPK ) abutment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient aged 18 - 80 yrs.
2. Implants treatment planned for single crown rehabilitation.
3. Submerged implant placement.
4. Patients willing to participate in a twelve month study.
5. Up to 2 implants per patient will be allowed.

Exclusion Criteria:

1. Active periodontal disease.
2. Systemic condition and medication that may affect soft and hard tissue healing.
3. Pregnancy or intention to become pregnant in the next twelve months.
4. Parafunctional occlusal scheme and habits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Soft tissue evaluation: | 12 month
  Three month following abutment connection (approximately 2 months following cementation of the final crowns) baseline measurement will be taken. This will include probing pockets depth (PPD) and bleeding on probing (BOP) dichotomized in to 0 and 1 This measurement will be repeated at 12 month post surgery.
Radiographic evaluation: | 12 month post surgery
  Bite wing radiographs will be used to assess changes in radiographic bone height.
  Baseline radiographs will be taking immediately following abutment connection and final radiographic evaluation will be taken 12 months post surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Maxillofacial Rehabillitaion School of Graduate Dentistry Rambam Health care campus, Haifa, Israel